CLINICAL TRIAL: NCT02385188
Title: Topical 5% Imiquimod Cream for Vulvar Paget's Disease: Clinical Efficacy, Safety and Immunological Response
Brief Title: Topical 5% Imiquimod Cream for Vulvar Paget's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Leiden University Medical Center (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); UMC Utrecht (Other); Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Joanne A. de Hullu, MD, PhD, MD PhD, University Medical Center Nijmegen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL51648.091.14
Record Dates: First submitted 2015-02-05; First posted 2015-03-11 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Paget Disease, Extramammary
Keywords: Extramammary Paget's disease; Vulva; Genital, female; imiquimod
MeSH Terms: conditions — Paget Disease, Extramammary | interventions — Imiquimod; Acetaminophen; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imiquimod (Experimental): Topical 5% imiquimod cream will be applicated to the vulvar skin lesion 3 times a week during 16 weeks.
  Interventions: Drug: Imiquimod; Drug: paracetamol; Drug: lidocaine in Vaseline ointment

INTERVENTIONS:
Drug: Imiquimod — topical 5% imiquimod cream 3 times a week for 16 weeks.
  Other Names: Aldara
Drug: paracetamol
Drug: lidocaine in Vaseline ointment

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and immunological response of topical 5% imiquimod cream for non-invasive vulvar Paget's disease.

DETAILED DESCRIPTION:
Vulvar Paget's disease is a rare skin tumour and generally seen in postmenopausal, Caucasian women as an erythematous, eczematous, scaling or ulcerating plaque. Initial symptoms are irritation, burning, pain and a skin lesion. The origin of vulvar Paget's disease is not yet entirely understood. The treatment of choice is surgical excision, despite high recurrence rates. The mutilating consequences of surgery can lead to impressive morbidity to address this, several series report the use of topical 5% imiquimod cream for vulvar Paget's disease.

The objective of this study is to assess the efficacy, evaluate the safety, immunological effect of topical 5% imiquimod cream for vulvar Paget's disease and the quality of life during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-invasive vulvar Paget's disease, primary or recurrence after earlier surgery;
* Willing and able to comply with the protocol and to provide informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

* Invasive vulvar Paget's disease;
* Underlying adenocarcinoma;
* Treatment of the vulva with topical 5% imiquimod cream during the last 6 months;
* Participation in a study with another investigational product within 30 days prior to enrolment in this study;
* Hypersensitivity to any component of topical 5% imiquimod cream (methylhydroxybenzoate (E218), propylhydroxybenzoate (E216), cetylalcohol, atearylalcohol);
* Patients with autoimmune disorders;
* Immune compromised patients (e.g. HIV patients, patients with a history of transplantation);
* Insufficient understanding of the Dutch or English language;
* Pregnant women;
* Lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Clinical response | 12 weeks after the end of treatment
  Clinical response will be assessed by vulvar examination and measurement and is defined as complete remission, partial remission (decrease by ≥50% of total lesion size) or no remission.

SECONDARY OUTCOMES:
Tolerability questionnaire | 4, 10 and 16 weeks after the start of treatment
  Tolerability will be assessed in a descriptive manner with a tolerability questionnaire with the following questions:
  1. Have you used paracetamol during treatment?
     1. How many days?
     2. What dosage?
     3. Was the use sufficient?
  2. Have you used lidocaine in Vaseline ointment during treatment?
     1. How many days?
     2. What dosage?
     3. Was the use sufficient?
  3. Have you stopped the treatment with imiquimod because of side effects/pain?
Adverse events | 4, 10 and 16 weeks after the start of treatment
  Most common adverse events will be evaluated with the following questions:
  1. Have you been nauseous? No / a little (less than 3 days per week) / severe (more than 3 days a week) / Yes, daily.
  2. Have you had a head ache? No / a little (less than 3 days per week) / severe (more than 3 days a week) / Yes, daily.
  3. Have you felt more tired than you normally are? No / a little (less than 3 days per week) / severe (more than 3 days a week) / Yes, daily.
Immunological response | Baseline, 4 and 28 weeks after start of treatment
  Vulvar skin biopsies will be taken at baseline, 4 and 28 weeks after the start of
Quality of life: general. | Baseline, 4 and 28 weeks after start of treatment.
  The questionnaire EQ5D (EuroQOL 5 Dimensions questionnaire) will be used.
Quality of life: dermatology specific. | Baseline, 4 and 28 weeks after start of treatment.
  The questionnaire DLQI (Dermatology Life Quality Index) will be used.
Quality of life: sexuality. | Baseline, 4 and 28 weeks after start of treatment.
  The questionnaire FSDS (Female Sexual Distress Scale) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne de Hullu, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (7):
- Netherlands (7):
  - Netherlands Cancer Institute, Amsterdam
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboudumc, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- [Derived] van der Linden M, van Hees CL, van Beurden M, Bulten J, van Dorst EB, Esajas MD, Meeuwis KA, Boll D, van Poelgeest MI, de Hullu JA. The Paget Trial: topical 5% imiquimod cream for noninvasive vulvar Paget disease. Am J Obstet Gynecol. 2022 Aug;227(2):250.e1-250.e8. doi: 10.1016/j.ajog.2022.04.012. Epub 2022 Apr 18. PMID 35447145
- [Derived] van der Linden M, Meeuwis K, van Hees C, van Dorst E, Bulten J, Bosse T, IntHout J, Boll D, Slangen B, van Seters M, van Beurden M, van Poelgeest M, de Hullu J. The Paget Trial: A Multicenter, Observational Cohort Intervention Study for the Clinical Efficacy, Safety, and Immunological Response of Topical 5% Imiquimod Cream for Vulvar Paget Disease. JMIR Res Protoc. 2017 Sep 6;6(9):e178. doi: 10.2196/resprot.7503. PMID 28877863